CLINICAL TRIAL: NCT01703754
Title: A Phase II Randomized, Open Label Study of Ad-RTS-hIL-12 Monotherapy or Combination With Palifosfamide in Subjects With Recurrent/Metastatic Breast Cancer and Accessible Lesions
Brief Title: Adenoviral Vector Monotherapy or Combination With Chemotherapy in Subjects With Recurrent/Metastatic Breast Cancer.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After SRC review and Sponsor's halting palifosfamide development, data was collected for Part 1, Arm A. Doses of 80, 100, and 140 mg were used. The SRC reduced 140 mg to 100 mg, then to 80 mg. The study ended with one subject enrolled at 80 mg daily.
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATI001-201
Record Dates: First submitted 2012-08-29; First posted 2012-10-10 (Estimated); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Nos Metastatic Recurrent
Keywords: Genetically Modified Organism; Metastatic Breast Cancer; Recurrent Breast Cancer; Breast Cancer; Palifosfamide; INXN1001; INXN2001; Adenoviral vector
MeSH Terms: conditions — Breast Neoplasms | interventions — veledimex; isophosphamide mustard; Palivizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ad-RTS-hIL-12 and veledimex (Experimental): Experimental study drug monotherapy arm (A)
  Interventions: Genetic: Ad-RTS-hIL-12 and Veledimex
- Ad-RTS-hIL-12 and Palifosfamide (Experimental): Study drug combination therapy arm (C)
  Interventions: Genetic: Ad-RTS-hIL-12 and Veledimex; Drug: Palifosfamide

INTERVENTIONS:
Genetic: Ad-RTS-hIL-12 and Veledimex — Oral activator ligand with adenoviral vector injection of cancer lesions
  Other Names: Adenoviral Vector; Oral activator ligand
Drug: Palifosfamide — Small molecule chemotherapy, IV administration
  Other Names: Pali
  Arms: Ad-RTS-hIL-12 and Palifosfamide

SUMMARY:
Phase II, randomized, safety and efficacy study in recurrent/metastatic breast cancer with accessible lesions.

Primary End point is rate of Progression Free Survival (PFS) at the 16 week treatment time point. Hypothesis: Adenoviral vector (Ad-RTS-hIL-12) alone and in combination with chemotherapy (palifosfamide) is safe and efficacious.

DETAILED DESCRIPTION:
Multicenter, open-label, randomized study evaluating the safety and efficacy of INXN-1001 (veledimex) and INXN-2001 (Ad-RTS-hIL-12) alone and in combination with palifosfamide.

Part 1 is the safety run-in where a safety assessment will be made after 1 cycle of therapy.

Part 2, eligible subjects will be randomly assigned to active treatment Arms A or C.

Once the monotherapy (Arm A) is determined to be safe and tolerable, Part 1 combination therapy (Arm C) will begin.

Subjects should receive six cycles of study treatment, in the absence of meeting withdrawal criteria.

ELIGIBILITY:
Inclusion criteria:

1. Males or females ≥ 18 years of age
2. Histologically or cytologically confirmed adenocarcinoma of the breast, either locally recurrent or metastatic disease with injectable lesions, for which no proven curative therapy exists.
3. Failed or progressed on at least 1 prior systemic chemotherapy regimen ± biologic/experimental therapy (if first-line therapy, failure or progression during the first 30 days).
4. Resolution of all treatment-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy ≤ Grade 2 and alopecia.
5. A minimum of 2 lesion(s) assessed by imaging using mRECIST v1.1.
6. Eastern Cooperative Oncology Group performance status 0, 1, 2
7. Male and female subjects must agree to use a highly reliable method of birth control.
8. Adequate bone marrow reserve as indicated by:

   1. Absolute neutrophil count > 1500/μL (without use of growth factors within 7 days)
   2. Absolute lymphocyte count > 700/μL (without use of growth factors within 7 days)
   3. Platelet count > 100,000/mm3 (without transfusion in prior 7 days)
   4. Hemoglobin > 9.0 g/dL (without transfusion in prior 7 days)
9. Estimated glomerular filtration rate using the Modification of Diet in Renal Disease equation: eGFR ≥ 60 mL/min/1.73 m2
10. Adequate liver function as evidenced by the following:

    1. Bilirubin ≤ 1.5 times the upper limits of normal (ULN)
    2. Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤ 2.5×ULN, in the case of liver metastases ≤ 5×ULN

Exclusion Criteria:

1. Subjects with human epidermal growth factor receptor 2 (HER2)/neu-positive (immunohistochemistry [IHC]) 3+ or fluorescence in situ hybridization-amplified) breast tumors who are eligible for, but who have not received HER2-targeted therapy (eg, trastuzumab)
2. Concomitant anticancer therapies
3. Prior therapies discontinuation periods:

   1. Radiation within 3 weeks of enrollment
   2. Chemotherapy within 4 weeks of enrollment
   3. Nitrosoureas within 6 weeks of enrollment
   4. Biologic therapy and/or immunomodulatory therapy, checkpoint inhibitors within 6 weeks of enrollment
   5. No washout period is required for endocrine therapy
4. Radiation therapy encompassing >25% of bone marrow
5. History of bone marrow or stem cell transplantation
6. Any congenital or acquired condition leading to inability to generate an immune response
7. Immunosuppressive therapy:

   1. Systemic immunosuppressive drugs including corticosteroids (prednisone equivalent >10 mg/day)
   2. Immune suppression/requiring immunosuppressive drugs, including organ allografts
   3. Active autoimmune disease requiring the equivalent of >10 mg/day of prednisone
8. Major surgery within 4 weeks of study treatment
9. History of prior malignancy, unless the prior malignancy was diagnosed and definitively treated ≥5 years previously with no subsequent evidence of recurrence
10. Subjects with brain or subdural metastases, unless local therapy has completed and corticosteroids have been discontinued for this indication for ≥4 weeks before starting study treatment.
11. Any medications that induce, inhibit, or are substrates of cytochrome P450 (CYP450) 3A4 within 7 days prior to the first dose of study drug
12. Subjects with meningeal carcinomatosis
13. Known significant hypersensitivity to study drugs or excipients
14. History of malabsorption syndrome or other condition that would interfere with enteral absorption
15. International Normalized Ratio (INR) and activated partial thromboplastin time [PTT] <1.5 x ULN, if not therapeutically anticoagulated.
16. New York Heart Association (NYHA) Class II or greater congestive heart failure OR active ventricular arrhythmia requiring medication
17. Any other unstable or clinically significant concurrent medical condition
18. Localized infection at site of injectable lesion(s) requiring antiinfective therapy within 2 weeks of the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2014-08-07 (Actual); Study Completion 2014-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaymes Holland, Study Director — Alaunos Therapeutics
Locations (8):
- United States (8):
  - Baptist Cancer Institute, Jacksonville, Florida
  - Henry Ford Health System, Detroit, Michigan
  - Billings Clinic, Billings, Montana
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Greenville Hospital System, Greenville, South Carolina
  - The Jones Clinic, PC, Germantown, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Evergreen Hematology & Oncology, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following the decision by the SRC the study will only collect data for the part 1, arm A group. Three dose level cohorts (140 mg, 100 mg, 80 mg) for INXN-1001 are used instead of the original single INXN-1001 dose level.
  Summaries that were based on part and treatment arm will instead be by dosage level of INXN-1001 where appropriate, with an overall group containing data from all dosage levels.
Groups:
- Ad-RTS-hIL-12 + Veledimex 140 mg: Ad-RTS-hIL-12 by intratumoral injection + Veledimex 140 mg daily for 7 days every 21-day cycle
- Ad-RTS-hIL-12 + Veledimex 100 mg Daily: Ad-RTS-hIL-12 by intratumoral injection + Veledimex 100 mg daily for 7 days every 21-day cycle
- Ad-RTS-hIL-12 + Veledimex 80 mg Daily: Ad-RTS-hIL-12 by intratumoral injection + Veledimex 80mg daily for 7 days every 21-day cycle
Period: Overall Study
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Started | 7 | 4 | 1
Completed (Completed 6 cycles of treatment) | 2 | 1 | 0
Not Completed | 5 | 3 | 1
Not completed — Clinically significant disease progression | 2 | 2 | 1
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population is defined as all subjects who receive at least one dose of study treatment (veledemix capsule and/or an injection of Ad-RTS-hIL-12).
Groups:
- Total: Total of all reporting groups
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily | Total
Number analyzed (Participants) | 7 | 4 | 1 | 12
Age, Continuous [Median (Full Range); unit: years] | 65.0 [38 to 88] | 58.0 [51 to 74] | 61.0 [61 to 61] | 62.5 [38 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 1 | 11
  Male | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 4 | 1 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 4 | 3 | 1 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 161.8 (8.72) | 163.8 (8.84) | 147.3 (0) | 161.3 (9.11)
Weight [Mean (Standard Deviation); unit: kg] | 62.50 (13.498) | 71.15 (17.731) | 59.00 (0) | 65.09 (14.357)
BMI [Mean (Standard Deviation); unit: kg/m2] | 23.875 (4.7718) | 26.306 (5.1260) | 27.192 (0) | 24.962 (4.6311)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: This measure will capture the incidence of Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and AEs leading to discontinuation. As per the protocol, safety and tolerability were assessed by monitoring adverse events, physical examinations, vital signs, electrocardiograms (ECGs), and clinical laboratory evaluations.
Time Frame: 16 months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 7 | 4 | 1
participants
  Any TEAE | 7 | 4 | 1
  Treatment-related TEAE | 7 | 4 | 1
  Grade 3 or higher TEAE | 6 | 2 | 1
  Treatment-related Grade 3 or higher TEAE | 5 | 2 | 1
  TEAE leading to death | 0 | 0 | 1
  Serious TEAE | 3 | 2 | 1
  TEAE leading to discontinuation | 2 | 2 | 1

2. Primary Outcome: 16-Week Progression-Free Survival (PFS) Rate
Description: This is the primary efficacy endpoint, defined as the proportion of subjects who had not progressed or died prior to 16 weeks from the date of their first dose. Progression was determined by modified Response Evaluation Criteria in Solid Tumors
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 7 | 4 | 1
participants | 2 | 1 | 0

3. Secondary Outcome: Best Overall Response (BOR) by mRECIST v1.1
Description: Best Overall Response (BOR) was determined for each evaluable subject up to their final tumor assessment. Per the modified Response Evaluation Criteria in Solid Tumors (mRECIST) v1.1, responses were defined as: Complete Response (CR), disappearance of all non-nodal target lesions and reduction in short axis of pathological lymph nodes to <10 mm; Partial Response (PR), at least a 30% decrease in the sum of diameters of target lesions from baseline; Progressive Disease (PD), at least a 20% increase in the sum of diameters from the smallest sum recorded; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD
Time Frame: 24 weeks
Population: The Efficacy Evaluable population is defined as all subjects who receive at least one dose of study treatment (veledimex capsule and/or an injection of Ad-RTS-hIL-12) and have at least one post-screening mRECIST response evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 4 | 3 | 1
Participants
  Best objective response of stable disease (SD) | 2 | 1 | 0
  Best objective response of unequivocal progression (UPD) | 2 | 2 | 1

4. Secondary Outcome: Estimate PFS by Modified RECIST v1.1
Description: Progression-free survival (PFS) is the time in days from the first dose of study treatment to the first assessment on which the response is reported as disease progression or death due to any cause (whichever is first) + 1 day. Subjects withdrawing from the study will be censored at their last non-progressive disease response assessment. If a subject does not have a disease response assessment, the subject will be censored on the date of the first treatment as described above.
  Kaplan-Meier plots will not be presented; PFS will be listed only.
Time Frame: 16 months
Population: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 4 | 3 | 1
Days | 94 [1 to 113] | 64 [1 to 174] | 1 [1 to 1]

5. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From 0 to 24 Hours (AUC0-24) of INXN-1001
Description: The area under the plasma concentration versus time curve from time 0 to 24 hours (AUC0-24) for INXN-1001
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 7
Population: The PK population includes all subjects in the Safety Run-in (Part 1) who had sufficient plasma concentration data to derive the specified parameter. The number of participants analyzed may be less than the total number in the arm due to missed PK sample collections or samples of insufficient quality for analysis
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 7 | 4 | 1
ng*h/mL
  AUC0-24 (ng*h/mL) at C1D1 | 8103 (5200) | 5935 (2660) | 13350 (0)
  AUC0-24 (ng*h/mL) at C1D7: number analyzed (Participants) | 3 | 2 | 1
  AUC0-24 (ng*h/mL) at C1D7 | 19478 (2353) | 10334 (654) | 8604 (0)
  Dose-normalized m2/mg AUC0-24 (ng*h/mL) at C1D1 | 89.0 (36.1) | 105 (16) | 266 (0)
  Dose-normalized m2/mg AUC0-24 (ng*h/mL) at C1D7: number analyzed (Participants) | 3 | 2 | 1
  Dose-normalized m2/mg AUC0-24 (ng*h/mL) at C1D7 | 250.1 (101.4) | 193 (74) | 171 (0)

6. Secondary Outcome: Change From Baseline in MUC-1 Specific T-Cell Response by ELISPOT Assay
Description: To assess for a cellular immune response, the number of MUC-1 specific interferon-gamma (IFN-γ) secreting T-cells was measured from peripheral blood mononuclear cells (PBMCs) using an ELISPOT assay. Results are reported as spot-forming cells (SFC) per million PBMCs
Time Frame: Screening and the Post-Treatment Safety Assessment visit (28 days after the last dose of study drug), with the final assessment occurring up to 7 months after the start of treatment.
Population: The Efficacy Evaluable population included all subjects who received at least one dose of study treatment and had at least one post-screening mRECIST response evaluation. The number of participants analyzed for this specific biomarker may be less than the total number in the arm due to missed sample collections or samples of insufficient quality for analysis.
Measure: Mean (Standard Deviation); unit: SFC/million PMBCs
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 7 | 4 | 1
SFC/million PMBCs
  Screening: Granzyme B ELISPOT Muc-1 (SFC/million PMBCs): number analyzed (Participants) | 6 | 4 | 1
  Screening: Granzyme B ELISPOT Muc-1 (SFC/million PMBCs) | 35.17 (0) | 0 (0) | 0 (0)
  Post-treatment Safety Assessment: Granzyme B ELISPOT Muc-1 (SFC/million PMBCs): number analyzed (Participants) | 5 | 2 | 1
  Post-treatment Safety Assessment: Granzyme B ELISPOT Muc-1 (SFC/million PMBCs) | 78.20 (75.16) | 30 (42.43) | 0 (0)

7. Secondary Outcome: Change From Baseline in Serum Interferon-gamma (IFN-γ) Levels
Description: Serum levels of IFN-γ were measured by immunoassay to assess the pharmacodynamic effect of the treatment
Time Frame: Screening, 24 hours after the first injection (Day 2), and at the Post-Treatment Safety Assessment visit, with the final assessment occurring up to 7 months after the start of treatment.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 7 | 4 | 1
pg/mL
  Screening: IFN-gamma (pg/mL) | NA (NA) — Below limit of quantitation (8.0 pg/mL) for all subjects | NA (NA) — Below limit of quantitation (8.0 pg/mL) for all subjects | NA (NA) — Below limit of quantitation (8.0 pg/mL) for all subjects
  Peak level in C1: IFN-gamma (pg/mL) | 354.84 (329.37) | 309.4 (358.37) | 68.1 (0)
  Post-treatment Safety Assessment: IFN-gamma (pg/mL) | NA (NA) — Below limit of quantitation (8.0 pg/mL) for all subjects | NA (NA) — Below limit of quantitation (8.0 pg/mL) for all subjects | NA (NA) — Below limit of quantitation (8.0 pg/mL) for all subjects

8. Secondary Outcome: Change From Baseline in Serum Interleukin-12 (IL-12) Levels
Description: Serum levels of IL-12 were measured by immunoassay to assess the pharmacodynamic effect of the treatment
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 7 | 4 | 1
pg/mL
  Screening:Interleukin-12(pg/mL) | 0.513 (0.409) | 0.485 (0.341) | 1.25 (0)
  Peak level in C1:IL-12 (pg/mL) | 33.8 (7.21) | 45.485 (15.264) | 47.7 (0)
  Post-treatment Safety Assessment:Interleukin-12 (pg/mL): number analyzed (Participants) | 6 | 3 | 1
  Post-treatment Safety Assessment:Interleukin-12 (pg/mL) | 0.81 (0.854) | 1.38 (1.67) | 2.1 (0)

9. Secondary Outcome: Change From Baseline in CD3+ CD4+ T-Cell Count
Description: Absolute counts of CD3+ CD4+ helper T-cells in peripheral blood were measured by flow cytometry to evaluate changes in immune cell populations.
Time Frame: Screening, Cycle 1 the Post-Treatment Safety Assessment visit Day 28 ± 3, and Follow-Up Tumor Assessment visits Day 63 ± 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cell/mcL
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 7 | 4 | 1
cell/mcL
  Screening: CD3+CD4+ (cell/mcL): number analyzed (Participants) | 2 | 3 | 1
  Screening: CD3+CD4+ (cell/mcL) | 845 (294.156) | 204.33 (82.59) | 263 (0)
  Post-treatment Safety Assessment::CD3+ CD4+(cell/mcL): number analyzed (Participants) | 4 | 2 | 1
  Post-treatment Safety Assessment::CD3+ CD4+(cell/mcL) | 337.75 (155.513) | 218.00 (114.55) | 104 (0)
  Follow-up Tumor Assessment: CD3+CD4+ (cell/mcL): number analyzed (Participants) | 3 | 1 | 0
  Follow-up Tumor Assessment: CD3+CD4+ (cell/mcL) | 367.33 (75.80) | 290 (0) |

10. Secondary Outcome: Change From Baseline in CD3+ CD8+ T-Cell Count
Description: Absolute counts of CD3+ CD8+ cytotoxic T-cells in peripheral blood were measured by flow cytometry to evaluate changes in immune cell populations
Time Frame: as for outcome 9
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cell/mcL
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 7 | 4 | 1
cell/mcL
  Screening: CD3+CD8+ (cell/mcL): number analyzed (Participants) | 2 | 3 | 1
  Screening: CD3+CD8+ (cell/mcL) | 1021 (702.86) | 168 (87.88) | 558 (0)
  Post-treatment Safety Assessment: CD3+CD8+ (cell/mcL): number analyzed (Participants) | 4 | 2 | 1
  Post-treatment Safety Assessment: CD3+CD8+ (cell/mcL) | 500.75 (594.91) | 252.5 (106.77) | 159 (0)
  Follow-up Tumor Assessment: CD3+CD8+ (cell/mcL): number analyzed (Participants) | 3 | 1 | 0
  Follow-up Tumor Assessment: CD3+CD8+ (cell/mcL) | 527.67 (441.00) | 150 (0) |

11. Secondary Outcome: Maximum Plasma Concentration (Cmax) of INXN-1001
Description: The maximum observed plasma concentration (Cmax) of INXN-1001 following oral administration.
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 7. On Day 1, samples were collected pre-dose and at 0.5, 1, 2, 4, and 6 hours post-dose. On Day 7, samples were collected pre-dose and at 1-2 and 4-6 hours post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 7 | 4 | 1
ng/mL
  Cmax (ng/mL) at C1D1 | 1024 (705) | 536 (218) | 1130 (0)
  Cmax (ng/mL) at C1D7: number analyzed (Participants) | 3 | 2 | 1
  Cmax (ng/mL) at C1D7 | 1403 (55) | 706 (81) | 749 (0)
  Dose-normalized m2/mg Cmax (ng/mL) at C1D1 | 11.1 (5.5) | 9.7 (2.6) | 22.5 (0)
  Dose-normalized m2/mg Cmax (ng/mL) at C1D7: number analyzed (Participants) | 3 | 2 | 1
  Dose-normalized m2/mg Cmax (ng/mL) at C1D7 | 17.8 (6.3) | 13 (4) | 14.9 (0)
  C24h (ng/mL) at C1D1 | 73.9 (54.0) | 39.7 (15.5) | 72 (0)
  C24 (ng/mL) at C1D7: number analyzed (Participants) | 3 | 2 | 1
  C24 (ng/mL) at C1D7 | 251 (48.4) | 101 (28) | 99 (0)

12. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of INXN-1001
Description: The time to reach the maximum observed plasma concentration (Tmax) of INXN-1001 following oral administration
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 7
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 7 | 4 | 1
hours
  Tmax (h) at C1D1 | 3.7 (1.4) | 4.8 (2.5) | 4 (0)
  Tmax (h) at C1D7: number analyzed (Participants) | 3 | 2 | 1
  Tmax (h) at C1D7 | 3.3 (1.2) | 3.0 (2) | 1 (0)

13. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate (CBR) was a pre-specified secondary endpoint defined as the proportion of subjects with a best overall response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD), as assessed by modified RECIST (mRECIST) v1.1.
Time Frame: From the first dose of study treatment for up to 1 year.
Population: The protocol pre-specified that the Clinical Benefit Rate (CBR) would be calculated. However, the final Statistical Analysis Plan states that due to the study's early termination and small sample size, this rate was not calculated. Best Overall Response for each individual subject was determined and is reported in a separate outcome measure.
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 months
Arm/Group | Ad-RTS-hIL-12 + Veledimex 140 mg | Ad-RTS-hIL-12 + Veledimex 100 mg Daily | Ad-RTS-hIL-12 + Veledimex 80 mg Daily
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4 | 1/1
Serious Adverse Events (participants affected / at risk) | 4/7 | 2/4 | 1/1
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ad-RTS-hIL-12 + Veledimex 140 mg (N=7) | Ad-RTS-hIL-12 + Veledimex 100 mg Daily (N=4) | Ad-RTS-hIL-12 + Veledimex 80 mg Daily (N=1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ad-RTS-hIL-12 + Veledimex 140 mg (N=7) | Ad-RTS-hIL-12 + Veledimex 100 mg Daily (N=4) | Ad-RTS-hIL-12 + Veledimex 80 mg Daily (N=1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (4) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (6) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (9) | 3 (3) | 0 (0)
Fatigue (General disorders) | 4 (8) | 3 (3) | 1 (1)
Chills (General disorders) | 5 (7) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2) | 0 (0)
Local swelling (General disorders) | 1 (1) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Asthena (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema mucosal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (4) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Blood urea decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 1 (2) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Blood chloride increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Mylagia (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2013-06-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT01703754/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT01703754/SAP_001.pdf